CLINICAL TRIAL: NCT06675929
Title: Safety, Tolerability and Pharmacodynamics of BI 770371 Administered Intravenously in Patients With Compensated Cirrhosis Due to MASH: a Phase IIa, Multi-center, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: A Study to Test How Well BI 770371 is Tolerated by People With Cirrhosis Caused by a Liver Disease Called MASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1501-0004; U1111-1307-2105 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Compensated Liver Cirrhosis; Metabolic Dysfunction Associated Steatohepatitis (MASH)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 770371 (Experimental)
  Interventions: Drug: BI 770371
- Placebo for BI 770371 (Placebo Comparator)
  Interventions: Drug: Placebo for BI 770371

INTERVENTIONS:
Drug: BI 770371 — BI 770371
  Arms: BI 770371
Drug: Placebo for BI 770371 — Placebo for BI 770371
  Arms: Placebo for BI 770371

SUMMARY:
This study is open to people with cirrhosis caused by a liver disease called MASH (metabolic dysfunction-associated steatohepatitis). The purpose of this study is to find out how well a medicine called BI 770371 is tolerated.

Participants are put into 2 groups by chance. One group gets BI 770371 as an infusion into a vein and the other group gets placebo as an infusion into a vein. Placebo infusions look like BI 770371 infusions but do not contain any medicine. Participants get an infusion every 3 weeks for 12 weeks.

Participants are in the study for about 5 months. During this time, they visit the study site 16 times. This also includes 1 overnight stay at the study site. The doctors regularly check participants' health and collect information on any health problems of the participants. The results are compared between the 2 groups.

ELIGIBILITY:
Inclusion criteria

* ≥18 to ≤75 years old
* Male or female participants
* Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of use is provided in the participant information
* Men able to father a child must be willing to use male contraception (condom or sexual abstinence) consistently and correctly until end of study. A list of contraception methods meeting these criteria and instructions on the duration of use is provided in the participant information
* Signed and dated written informed consent in accordance with ICH-Good Clinical Practice (GCP) and local legislation prior to admission to the trial
* Patients meeting criteria for Child-Pugh category A
* Adequate organ function or liver laboratory tests defined as all of the following:

  * Total bilirubin ≤1.5 mg/dL. If the total bilirubin is > upper limit of normal (ULN) and a ≤1.5 mg/dL, the direct bilirubin must be <50% of total bilirubin
  * For patients with Gilbert's syndrome: total bilirubin ≤3x ULN or direct bilirubin ≤1.5x ULN
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤5x ULN
  * Alkaline Phosphatase <1.5x ULN
  * International Normalized Ratio (INR) ≤1.4
  * Model for End-Stage Liver Disease (MELD) score <12
  * Platelet count ≥110 000/mL
  * Albumin >3.4 g/dl

Exclusion criteria

* Major surgery (major according to the investigator's assessment) performed within 24-weeks prior to randomization, major surgery planned within 6 months after screening (e.g. hip replacement), or bariatric surgery within 2 years prior to randomization
* Any documented active or suspected malignancy or history of malignancy within 5-years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix. Specifically, any patients with suspected, confirmed, or history of hepatocellular carcinoma will be excluded
* Suspected or confirmed portal vein thrombosis within 6 months of enrollment
* History of liver transplantation
* Current listing for liver transplantation
* Present or past evidence of hepatic decompensation, in the opinion of the investigator, including but not limited to variceal hemorrhage, ascites, and/or hepatic encephalopathy
* Patients with clinically significant portal hypertension defined by any one of the following:

  * FibroScan ≥25 Kilo Pascal (kPA) if the platelets are ≥150,000/μL
  * FibroScan ≥20 kPA if platelets are <150,000/μL
  * Evidence of esophageal or gastric varices (≥grade1) on the most recent endoscopy
  * Enhanced liver fibrosis (ELF) ≥11.3
  * Hepatic venous pressure gradient (HVPG) ≥10 mm Hg
* further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent, drug-related adverse events in the BI 770371 and placebo arms | Up to Week 15

SECONDARY OUTCOMES:
Occurrence of adverse events (including clinically relevant findings from medical examination, safety laboratory tests, 12-lead ECG, vital signs, and assessment of local tolerability | Up to Week 22
Change from baseline in the fibrosis-related soluble biomarker PRO-C3 after 12 weeks of treatment | Baseline , at Week 12
  PRO = propeptide

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - The Institute for Liver Health II dba Arizona Clinical Trials, Chandler, Arizona
  - Southern California Research Center, Coronado, California
  - Catalina Research Institute, LLC-Montclair-49051, Montclair, California
  - Knowledge Research Center, Orange, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Peak Gastroenterology Associates-Colorado Springs-67762, Colorado Springs, Colorado
  - Evolution Clinical Trials, Miami, Florida
  - Blessed Health Care, Miami, Florida
  - Progressive Medical Research, Port Orange, Florida
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Houston Research Institute, Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https:// www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'. For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com